CLINICAL TRIAL: NCT05066997
Title: A Phase 2/3 Double-Masked, Randomized, 2 Stage, Multicenter Study of the Efficacy and Safety of OCS-01 Eye Drops in Subjects With Diabetic Macular Edema
Brief Title: A Pivotal Safety and Efficacy Study of OCS-01 Eye Drops in Participants With Diabetic Macular Edema (DIAMOND 1)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oculis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX219
Record Dates: First submitted 2021-09-02; First posted 2021-10-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Macular Edema
Keywords: Topical ophthalmic suspension; Eye drop
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OCS-01 (Experimental): dexamethasone ophthalmic suspension,1.5% [15 mg/ mL]
  Interventions: Drug: Dexamethasone ophthalmic suspension (OCS-01)
- Vehicle Vehicle (Placebo Comparator): Placebo is a Vehicle ophthalmic suspension of OCS-01
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Dexamethasone ophthalmic suspension (OCS-01) — Stage 1: Participants will be dosed with one eye drop of OCS-01 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 6 weeks (maintenance phase).
  Stage 2: Participants will be dosed with one eye drop of OCS-01 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 46 weeks (maintenance phase).
  Other Names: Dexamethasone
  Arms: OCS-01
Drug: Vehicle — Stage 1: Participants will be dosed with one eye drop of vehicle 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 6 weeks (maintenance phase).
  Stage 2: Participant will be dosed with one eye drop of vehicle 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 46 weeks (maintenance phase).
  Other Names: Placebo
  Arms: Vehicle Vehicle

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of the topical ophthalmic administration of OCS- 01 as compared to Vehicle in participants with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
A Phase 2/3 Pivotal Double-masked, Randomized, Vehicle-controlled, 2 stage, Multicenter Study of the Efficacy and Safety of OCS-01 Eye Drops in Participants with Diabetic Macular Edema

Stage 1: To select a dose and dosing regimen for OCS-01 in participants with DME and evaluate the efficacy and safety of OCS-01 as compared to Vehicle in participants with DME.

Stage 2: To evaluate the efficacy and safety of OCS-01 as compared to Vehicle at Week 52 in participants with DME.

ELIGIBILITY:
Inclusion Criteria (selection) - Stage 1:

1. Have a signed informed consent form before any study-specific procedures are performed.
2. Have DME with presence of intraretinal and/or subretinal fluid in the study eye, with central subfield thickness (CST) of ≥310 µm by SD-OCT at screening (Visit 1) (as assessed by an independent reading center).
3. Have a documented diagnosis of type 1 or type 2 diabetes mellitus at Visit 1 (Screening).

Inclusion Criteria (selection) - Stage 2:

1. Have a signed informed consent form before any study-specific procedures are performed.
2. Have DME with presence of intraretinal and/or subretinal fluid in the study eye, with central subfield thickness (CST) of ≥310 µm by SD-OCT at screening (Visit 1) (as assessed by an independent reading center).
3. Have a documented diagnosis of type 1 or type 2 diabetes mellitus prior to Visit 1 (Screening).

Exclusion criteria (selection) - Stage 1 and Stage 2:

1. Have macular edema considered to be because of a cause other than DME.
2. Have a decrease in BCVA because of causes other than DME.
3. Have a known history of significant macular ischemia which would prevent gain in visual acuity in the study eye.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean Change in BCVA (Best Corrected Visual Acuity) | Week 52
  Assessed using ETDRS (Early Treatment Diabetes Retinopathy Study) letters score: higher numbers on the ETDRS chart representing better visual acuity

SECONDARY OUTCOMES:
Percentage of Participants with a 3-line or Greater Gain in BCVA | Baseline, Week 52
  BCVA will be assessed by ETDRS letters score: higher numbers on the ETDRS chart representing better visual acuity.
Mean Change in BCVA | Baseline, Week 12 and Week 24
  BCVA will be assessed using ETDRS letters score: higher numbers on the ETDRS chart representing better visual acuity.
Mean Change in Central Subfield Thickness (CST) | Baseline, Week 52
  CST will be measured by SD-OCT.

OTHER OUTCOMES:
Number of Participants With Treatment Emergent Adverse events (TEAEs) | Up to Week 52
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant. TEAEs are those AEs that occur after administration of the study product and are therefore temporally associated with the use of the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Veeral S Sheth, MD, Principal Investigator — University Retina - Lemont
Locations (52):
- United States (40):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Phoenix Retina Associates, Phoenix, Arizona
  - Retina Partners of Northwest Arkansas, Springdale, Arkansas
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retinal Consultants Medical Group, Modesto, California
  - California Eye Specialists Medical Group, Pasadena, California
  - California Eye Specialists Medical Group, Redlands, California
  - Retina Consultants of Southern California, Redlands, California
  - California Retina Consultants, Santa Maria, California
  - Retina Group Of New England, Waterford, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - Florida Retina Institute, Jacksonville, Florida
  - MedEye Associates, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Associates, Elmhurst, Illinois
  - University Retina, Lemont, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Retina-Vitreous Surgeons of Central New York, Liverpool, New York
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Velocity (Meridian) Clinical Research, Cincinnati, Ohio
  - Verum Research LLC, Eugene, Oregon
  - Vision Research Solutions in Philadelphia, Philadelphia, Pennsylvania
  - Retina Consultants of Charleston, Beaufort, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Consultants of Austin/Austin Research Center for Retina, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Valley Retina Institute PA d.b.a. Gulf Coast Eye Institute, McAllen, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
- Hong Kong (2):
  - HKU Eye Centre, Hong Kong
  - Chinese University of Hong Kong Eye Centre, Kowloon
- India (6):
  - Shivam Retina Clinic and Eye Hospital, Surat, Gujarat
  - Nethra Eye Hospital, Bengaluru, Karnataka
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Sarakshi Netralaya, Nagpur, Maharashtra
  - L V Prasad Eye Institute, Bhubaneswar, Odisha
  - ICARE Eye Hospital & Post Graduate Institute, Noida, Uttar Pradesh
- Taiwan (4):
  - Changhua Christian Hospital, Changhua, Changhua
  - China Medical University Hospital, Taichung, Taichung
  - Taipei Veterans General Hospital, Taipei, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District, Taoyuan

IPD SHARING:
Plan to Share IPD: No